CLINICAL TRIAL: NCT02712086
Title: Randomized Controlled Trial Prospective Single-center Open Evaluating the Efficacy of Supplementation (Adapted to the Post-operative Period) Current Protein After Bariatric Surgery Like Sleeve Gastrectomy
Brief Title: Controlled Trial Evaluating the Efficacy of Protein Supplementation in the Short Term After Bariatric Surgery
Acronym: PROTISLEEVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RECHMPL15_0173; UF 9590 (Other: Montpellier University Hospital)
Record Dates: First submitted 2016-03-14; First posted 2016-03-17 (Estimated); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- usual dietary management (No Intervention): Control group: usual dietary management Following the intervention, the stomach of patients underwent many changes
- care of with usual dietary protein supplementation (Experimental): Intervention group: Usual dietary management with protein supplementation (30g) in addition to the usual inputs
  Interventions: Other: protein supplementation

INTERVENTIONS:
Other: protein supplementation — Protein supplementation : Protein intake of 30 grams of protein in addition to the usual inputs (to the recommended amounts of 60 to 120 g per day), upon the resumption of oral intake until the fifth week after sleeve gastrectomy.
  Arms: care of with usual dietary protein supplementation

SUMMARY:
The main objective will be to evaluate the effect at 5 weeks of nutritional management associated with protein supplementation (adapted to the post-operative period) on the maintenance of lean body mass at the whole body in obese patients after a sleeve gastrectomy.

Secondary objectives will assess protein intake, food safety, the effect of protein supplementation on body fat in the entire body and the metabolic rate and the impact on quality of life and post-operative joint pain.

DETAILED DESCRIPTION:
The main objective will be to evaluate the effect at 5 weeks of nutritional management associated with protein supplementation (adapted to the post-operative period) on the maintenance of lean body mass at the whole body in obese patients after a sleeve gastrectomy.

Secondary objectives will assess protein intake, food safety, the effect of protein supplementation on body fat in the entire body and the metabolic rate and the impact on quality of life and post-operative joint pain.

There is still no study evaluating the protein supplementation adapted patients after sleeve gastrectomy on maintaining lean body mass.

ELIGIBILITY:
Inclusion Criteria:

* surgical management of sleeve gastrectomy kind

Exclusion Criteria:

* food allergies
* Weight> 135 kg (maximum weight supported by the DXA)
* orthopedic prosthesis (hip, knee ...) that would make it impossible to interpret the measurement of DXA
* History of bariatric surgery: adjustable gastric banding, vertical banded gastrectomy ...

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2016-10-19 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Changes in lean mass (kg) will be assessed at the level of whole-body dual-energy X-ray absorptiometry (DXA) | up to 1 month

SECONDARY OUTCOMES:
food diary | 5 weeks after the hospital discharge
  The actual protein intake will be assessed using a food diary over 5 weeks completed by the patient
change rate IGF1, IGFBP3 | up to 1 month
  change rate IGF1, IGFBP3 between hospitalization and 1 month of hospital discharge
the quality of life | up to 1 month
  The evolution of the quality of life will be assessed through a specific scale, Baros score.
the quality of life | up to 5 years
  The evolution of the quality of life will be assessed through a specific scale, Baros score.
change rate IGF1, IGFBP3 | up to 5 years
  change rate IGF1, IGFBP3 between hospitalization and 5 years follow up

CONTACTS AND LOCATIONS:
Overall Officials: David NOCCA, Principal Investigator — University Hospital, Montpellier
Locations (1):
- UHMontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Maimoun L, Aouinti S, Puech M, Lefebvre P, Deloze M, de Santa Barbara P, Renard E, Christol JP, Myzia J, Picot MC, Mariano-Goulart D, Nocca D. Changes in Lean Tissue Mass, Fat Mass, Biological Parameters and Resting Energy Expenditure over 24 Months Following Sleeve Gastrectomy. Nutrients. 2023 Feb 27;15(5):1201. doi: 10.3390/nu15051201. PMID 36904198
- [Result] Maimoun L, Aouinti S, Puech M, Lefebvre P, Humbert L, Deloze M, de Santa Barbara P, Maimoun-Nande L, Boudousq V, Cristol JP, Renard E, Picot MC, Mariano-Goulart D, Nocca D. Modification of bone architecture following sleeve gastrectomy: a five-year follow-up. J Bone Miner Res. 2025 Feb 2;40(2):251-261. doi: 10.1093/jbmr/zjae202. PMID 39693376